CLINICAL TRIAL: NCT02496871
Title: Remote Delivery of Weight Management by Phone and Social Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Blue Cross Blue Shield (Other); Kansas City Area Life Sciences Institute, Inc. (Other)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002758
Record Dates: First submitted 2015-06-30; First posted 2015-07-14 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Media Exposure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KWMP-GP (Active Comparator): Weekly group phone calls for 6 months. Group phone calls will last about 45 minutes each. Phone calls will include groups of 12-18 participants.
  Interventions: Behavioral: Group Phone Calls
- KWMP-SM (Experimental): Participants interact through a private Facebook group. New activities for participants to complete each week for 6 months.
  Interventions: Behavioral: Social Media

INTERVENTIONS:
Behavioral: Group Phone Calls — University of Kansas Weight Management Program - Group Phone calls
  Other Names: KWMP-GP
  Arms: KWMP-GP
Behavioral: Social Media — University of Kansas Weight Management Program - Social Media (Facebook)
  Other Names: KWMP-SM
  Arms: KWMP-SM

SUMMARY:
The purpose of this study is to compare two different weight management delivery methods, social media versus a traditional care model.

DETAILED DESCRIPTION:
Obesity is a major public health issue as 68% of the US population is either overweight or obese. Weight loss and weight loss maintenance is difficult. Traditionally, successful weight loss programs are weekly behaviorally-based clinics which utilize a combination of calorie restriction and physical activity. Traditional "face to face" weekly meetings may not be feasible for everyone.

An alternative to provide weight loss and weight maintenance created by KUMC researchers uses weekly group phone conference calls. While this method produced equal weight loss with fewer burdens to participants when compared to the traditional "face to face" format, weight regain during maintenance was still high.

This study will investigate a new delivery method (social media platform "Facebook") compared to the group phone conference calls. In the social media platform participants will be able to socialize with other participants in their group by commenting on posts from other participants or posting messages themselves. Social media delivered programs have potential to be a more a cost-effective approach to reach a large group of individuals.

Participants who are eligible and decided to be in this study will take part in study related activities for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 30 to 45 kg/m^2
* Have access to a computer, smart phone, or tablet
* Give informed consent to participate

Exclusion Criteria:

* Unable to participate in moderate intensity PA (i.e., walking)
* Participation in a weight loss or physical activity program in the previous 6 mos.
* Greater than 3, 30-min bouts of planned exercise/week
* Not weight stable (±4.6 kg) for 3 mos. prior to intake
* Unwilling to be randomized to 1 of the 2 study groups
* Report being pregnant during the previous 6 mos., currently lactating, or planned pregnancy in the following 6 mos.
* Serious medical risk such as cancer, recent cardiac event (i.e. heart attack, stroke, angioplasty) as determined by the individual's PCP via the clearance to participate in the investigation
* Current use of antipsychotics or untreated depression
* Adherence to specialized diet regimens, i.e., multiple food allergies, vegetarian, macrobiotic
* Binge eating disorder as assessed by the Binge Eating Scale
* Living in the same household as another study participant

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change in weight | Change from Baseline to Month 6

SECONDARY OUTCOMES:
Change in BMI | Change from Baseline to Month 6
Physical activity - steps | Month 6
  Measured using pedometer to report steps per day on a weekly basis
Physical activity - total minutes | Month 6
  Average of total minutes per week of physical activity
Physical activity - ActiGraph Activity Level (Count/Minute; CPM) | 7 days
  Average ActiGraph counts/minute over 7-day period. Activity level based on cut points used in NHANES as described by Troiano. Cut points used will be Sedentary: 0 - 99 CPM; Light: 100 - 2019 CPM; Moderate: 2020 - 5998 CPM; Vigorous: 5999 - ∞ CPM.
Dietary assessment - self-reported log | Month 6
  Participants will complete dietary intake log, including 2 weekdays and 1 weekend day, using MyFitnessPal application prior to baseline and month 6 visits.
Quality of Life Assessment (SF-36) | Change from Baseline to Month 6
  Measured using the Short Form 36 (SF-12) Health Survey.
Quality of Life - Weight Related | Change from Baseline to Month 6
  Measured using the SHIELD-WQ-9 Questionnaire
Feasibility of Interventions - adherence to protocol procedures | Month 6
  Participants adherence to diet, physical activity and attendance/participation in weight loss sessions.

OTHER OUTCOMES:
Cost Analysis of Interventions | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Willis EA, Szabo-Reed AN, Ptomey LT, Steger FL, Honas JJ, Al-Hihi EM, Lee R, Vansaghi L, Washburn RA, Donnelly JE. Distance learning strategies for weight management utilizing social media: A comparison of phone conference call versus social media platform. Rationale and design for a randomized study. Contemp Clin Trials. 2016 Mar;47:282-8. doi: 10.1016/j.cct.2016.02.005. Epub 2016 Feb 12. PMID 26883282